CLINICAL TRIAL: NCT03866499
Title: A Randomized, Double-blind, Positive Controlled Phase III Study to Evaluate the Efficacy and Safety of BPI-7711 Capsule in Locally Advanced or Recurrent/Metastatic Treatment-naïve Non-small Cell Lung Cancer Patients With EGFR Mutation
Brief Title: A Study of BPI-7711 Capsule in Non-small Cell Lung Cancer Patients
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Beta Pharma Shanghai (Industry)
Responsible Party: Sponsor
Organization: Beta Pharma, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BPI-7711301
Record Dates: First submitted 2019-03-05; First posted 2019-03-07 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-08

CONDITIONS: NSCLC
Keywords: EGFR mutation; EGFR TKI; NSCLC
MeSH Terms: interventions — rezivertinib; Gefitinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BPI-7711 (Experimental): 180 mg BPI-7711 capsule + 250mg gefitinib placebo tablet, QD
  Interventions: Drug: BPI-7711; Drug: Placebo Tablet
- Gefitinib (Active Comparator): 180 mg BPI-7711 placebo capsule + 250mg gefitinib tablet, QD
  Interventions: Drug: Gefitinib; Drug: Placebo capsule

INTERVENTIONS:
Drug: BPI-7711 — 180 mg, oral, QD
  Other Names: BPI-7711 capsule
  Arms: BPI-7711
Drug: Gefitinib — 250 mg, oral, QD
  Other Names: Iressa
  Arms: Gefitinib
Drug: Placebo Tablet — 250 mg gefitinib placebo tablet, QD
  Other Names: placebo
  Arms: BPI-7711
Drug: Placebo capsule — 180 mg BPI-7711 placebo capsule, QD
  Other Names: placebo
  Arms: Gefitinib

SUMMARY:
A randomized, double-blind, positive controlled phase III study to evaluate the efficacy and safety of BPI-7711 capsule in locally advanced or recurrent/metastatic treatment-naïve non-small cell lung cancer patients with EGFR mutation

DETAILED DESCRIPTION:
This is a Phase III clinical study, which aims to compare the efficacy and safety of BPI-7711 capsule and gefitinib tablet in the treatment of initially-treated patients with locally advanced or recurrent metastatic with EGFR mutation.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed non-small cell lung cancer.
* The ECOG score of performance status is 0-1.
* Locally advanced or recurrent metastatic NSCLC that has never received systemic treatment.
* According to RECIST1.1 criteria, there is at least 1 measurable lesion that has not been previously irradiated.
* Prior to enrollment, a central laboratory testing report has confirmed that the tumor has one of two common EGFR mutations positive that are sensitive to EGFR-TKI therapy, accompanied with or not accompanied with other EGFR mutation, with the exception of exon 20 insertion.

Exclusion Criteria:

* Previously received systemic treatment for locally advanced or recurrent metastatic cancer.
* Primary T790M mutation-positive patient.
* Previous interstitial lung disease, drug-induced interstitial lung disease, radiation pneumonia requiring hormonal therapy, or any clinically proven active interstitial lung disease.
* Known active infections such as hepatitis B, hepatitis C, and human immunodeficiency virus.
* Local radiation therapy is carried out within 1 week; more than 30% bone marrow radiation therapy or extensive radiation therapy is performed within 4 weeks.
* ≤ 4 weeks from major surgery or ≤ 2 weeks from minor surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 369 (Actual)
Dates: Start 2021-04-30 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | up to approximately 16 months
  Progression-free survival evaluated by Blinded Independent Center Review

SECONDARY OUTCOMES:
Progression-free survival | up to approximately 16 months
  Progression-free survival evaluated by investigators
Objective response rate | up to approximately 16 months
  Objective response rate
Best objective response | up to approximately 16 months
  Best objective response
Disease control rate | up to approximately 16 months
  Disease control rate
Duration of response | up to approximately 16 months
  Duration of response
Overall survival | up to approximately 30 months
  Overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Yuankai Shi, Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Locations (3):
- China (3):
  - Cancer Hospital Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Linyi Cancer Hospital, Linyi, Shandong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Shi Y, Guo Y, Li X, Wu L, Chen Z, Yang S, Bi M, Zhao Y, Yao W, Yu H, Wang K, Zhao W, Sun M, Zhang L, He Z, Lin Y, Shi J, Zhu B, Wang L, Pan Y, Shi H, Sun S, Wen M, Zhou R, Guo S, Han Z, Yi T, Zhang H, Cang S, Yu Z, Zhong D, Cui J, Fang J, Gao J, Li M, Ma R, Jiang M, Qin J, Shu Y, Ye F, Hu S, Li W, Lu H, Yang M, Yi S, Zhang Y, Fan Y, Ji H, Liu Z, Wang H, Zhou X, Zhang D, Peng J, Shen H, Gao F, Wang T, Zhou A. Rezivertinib versus gefitinib as first-line therapy for patients with EGFR-mutated locally advanced or metastatic non-small-cell lung cancer (REZOR): a multicentre, double-blind, randomised, phase 3 study. Lancet Respir Med. 2025 Apr;13(4):327-337. doi: 10.1016/S2213-2600(24)00417-X. Epub 2025 Feb 3. PMID 39914443